CLINICAL TRIAL: NCT02617550
Title: Evaluation of the Effect of 0.4 mg Nitroglycerin Spray After Pretreatment With Multiple Once Daily Oral Doses of 2.5 mg, 5 mg and 10 mg Vericiguat (BAY 1021189) Each Given Over 14 ± 3 Days on Safety, Tolerability and Blood Pressure in a Multi-center, Randomized, Placebo-controlled, Double-blind Group Comparison Study in Stable Coronary Artery Disease (CAD) Patients Aged 30 to 80 Years
Brief Title: Vericiguat Drug-drug Interaction With Nitroglycerin in Stable Coronary Artery Disease Patients
Acronym: VENICE
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 17849; 2015-001444-11 (EudraCT Number)
Record Dates: First submitted 2015-11-11; First posted 2015-12-01 (Estimated); Last update posted 2021-12-29 (Actual); Status verified 2021-12

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — vericiguat; Nitroglycerin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vericiguat + Nitroglycerin (Experimental): Co-administration of vericiguat and nitroglycerin
  Interventions: Drug: Vericiguat (BAY1021189); Drug: Nitroglycerin
- Placebo + Nitroglycerin (Placebo Comparator): Aministration of matching placebo and nitroglycerin.
  Interventions: Drug: Placebo; Drug: Nitroglycerin

INTERVENTIONS:
Drug: Vericiguat (BAY1021189) — Vericiguat up-titration from 2.5 mg to 10 mg in an interval of 14 +/- 3 days: 2.5 mg vericiguat for 14 +/-3 days given as 2 x 1.25 mg tablets followed by 5 mg vericiguat for 14 +/-3 days given as 1 x 5 mg tablet followed by 10 mg vericiguat for 14 +/-3 days given as 2 x 5 mg tablets
  Arms: Vericiguat + Nitroglycerin
Drug: Placebo — Placebo for 14 +/-3 days given as 1 or 2 tablets [o.d.].
  Arms: Placebo + Nitroglycerin
Drug: Nitroglycerin — 0.4 mg nitroglycerin spray administered at 2.5 hours before treatment (vericiguat [trough] or placebo) on day 12, day 26 and day 40 at 4 hours after treatment (vericiguat [peak] or placebo) on day 13, day 27 and day 41

SUMMARY:
This study is intended to investigate the effect of nitroglycerin on vericiguat in patients with stable coronary artery disease (CAD). Nitroglycerin is the standard therapy to treat acute crisis of angina. Thus there is a high likelihood of co-administration of both drugs in the target indication of vericiguat, worsening heart failure (HF). Therefore, it is important to investigate the safety and tolerability of vericiguat and nitroglycerin, which may be used as unprescribed on-demand treatment by patients with acute episodes of angina pectoris.

ELIGIBILITY:
Inclusion Criteria:

Patients with stable CAD defined by

* coronary artery stenosis in any of the 3 main coronary vessels > 50% documented by coronary angiography within last 36 months or history of myocardial infarction
* Age: 30 to 80 years
* Body mass index (BMI): above/equal 18.0 and below/equal 36.0 kg / m²
* Female subjects must be of non-childbearing potential

Exclusion Criteria:

* Intervention e.g. revascularization by percutaneous coronary intervention (PCI) and/or coronary artery bypass graft (CABG) during the last 3 months
* Progressive angina with symptoms of worsening of angina within the < 3 months
* History of recent (< 6 months prior to the first screening examination) myocardial infarction or unstable angina
* Symptomatic carotid stenosis, or transient ischemic attack or stroke within 3 months prior or patients with stroke at more than 3 months prior with significant residual neurologic involvement
* Insulin dependent diabetes mellitus
* Clinically relevant cardiac ischemia
* Clinical significant persistent ischemia
* Atrial fibrillation, pacemaker, defibrillator, atrial ventricular (AV)-block II and III
* Systolic blood pressure below 110 or above 160 mmHg
* Diastolic blood pressure above 100 mmHg
* Heart rate below 50 or above 100 beats / min
* Estimated glomerular filtration rate < 30 mL/min/1.73m2

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2015-11-18 (Actual); Primary Completion 2016-05-18 (Actual); Study Completion 2016-08-11 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events as measure of safety and tolerability | approximately 1 year

SECONDARY OUTCOMES:
Blood pressure | approximately 1 year
  Regular measurement of blood pressure (mmHg) in supine, sitting and standing position.
Heart rate | approximately 1 year
  Regular measurement of heart rate (bpm) in supine, sitting and standing position.

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (6):
- Germany (6):
  - Heidelberg, Baden-Wurttemberg
  - Bonn, North Rhine-Westphalia
  - Wuppertal, North Rhine-Westphalia
  - Erfurt, Thuringia
  - Berlin
  - Hamburg

REFERENCES:
- See also: Click here to find results for studies related to Bayer products. — http://clinicaltrials.bayer.com/